CLINICAL TRIAL: NCT01752881
Title: Immunogenicity and Safety of a Trivalent Inactivated Influenza Vaccine, Formulation 2012-2013, in Non-Elderly Adult and Elderly Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLU12T13A
Record Dates: First submitted 2012-12-17; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Immunogenicity
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdimFlu-S (Experimental)
  Interventions: Biological: Influenza vaccine (split virion, inactivated); Biological: AdimFlu-S

INTERVENTIONS:
Biological: Influenza vaccine (split virion, inactivated) — AdimFlu-S, Inactivated Influenza Vaccine Trivalent Types A and B (Split) Formulation 2012-2013
  Dosage: 0.5mL/per syringe
  Administration route: Intramuscular Injection, once
  Other Names: AdimFlu-S Influenza Vaccine
Biological: AdimFlu-S

SUMMARY:
The purpose of this study is to evaluate the antibody response to each of the three influenza vaccine strains included in the licensed seasonal flu vaccine, as measured by hemagglutination inhibition (HAI) at three weeks post immunization in non-elderly and elderly subjects in compliance with the requirements of the current European Union (EU) recommendations for the evaluation of the immunogenicity for a new formulation of a licensed flu vaccine (CPMP/BWP/214/96).

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females and aged ≥ 18 years;
* Willing and able to adhere to visit schedules and all study requirements;
* Subjects read and signed the study-specific informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Immunogenicity endpoint: Seroprotection rate | At 3 weeks after vaccination
  Seroprotection rate is defined as the proportion of subjects with HAI titer ≥ 1:40.
Immunogenicity endpoint: Seroconversion rate | At 3 weeks after vaccination
  The seroconversion is defined as the HAI titer of the post-vaccination serum is at least 1:40 for those who had a negative pre-vaccination HAI serum titer or a four-fold or greater increase in HAI titers in subjects who had a positive pre-vaccination HAI serum titer. The seropositive is defined as the HAI titer ≥ 1:10, and the seronegative is defined as HAI titer < 1:10.
Immunogenicity endpoint: Geometric mean folds increase in HAI titer | At 3 weeks after vaccination

SECONDARY OUTCOMES:
Safety: Reactogenicity events | 7 days after vaccination
  Reactogenicity events are pre-specified adverse events systematically recorded for 7 days after vaccination. The selection of the events to be collected systematically is based on events expected to occur with wild-type influenza infection including fever (≥38°C), runny nose or nasal congestion, cough, sore throat, headache, muscle aches, vomiting, nausea and malaise. Furthermore, the local (injection site) reactions will also be evaluated that include soreness/pain, swelling, redness, ecchymosis and limitation of arm motion.
Safety: Serious and non-serious adverse events | Through day 21 post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Jen Chang, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan